CLINICAL TRIAL: NCT04730479
Title: Ultrasound Prediction of Radial Arterial Catheterization Failure in Patients Undergoing Cardiac or Aortic Surgery: a Prospective Study
Brief Title: Echography to Predict Radial Artery Catheterization Failure (EPRAC)
Acronym: EPRAC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0091
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Cardiac and Aortic Surgery
Keywords: ultrasonography; radial artery catheterization; probabilistic model; adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In patients undergoing cardiac or aortic surgery, the placement of a radial KTA is sometimes difficult, the purpose of this study is to do an ultrasound in order to evaluate the diagnostic values of the internal diameter of the radial artery to predict the failure to install the radial KTA.

DETAILED DESCRIPTION:
The Arterial Catheter (KTA) enables continuous measurement of invasive blood pressure in patients with accurate and reliable hemodynamic monitoring. Radial Artery Catheterization is the currently recommended placement site.

In patients undergoing cardiac or aortic surgery, placement of a radial KTA is sometimes difficult, with a failure rate of around 15%. It is also a source of local complications and prolongation of the anesthetic duration.

There is no predictive diagnostic test for failed radial KTA placement in anesthesia.

Accurately predicting the failure of radial catheterization by echography will, in the future, make it possible to offer "at risk" patients an immediate catheterization in an other site as for example brachial site.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years old
* Be operated for a scheduled cardiac or aortic surgery
* Be able to complete all the visits and follow the study procedures
* Subjects must be covered by public health insurance

Exclusion Criteria:

* Patients protected by law or Absence of signed informed consent
* Emergency Surgery Patient
* Patient already with an arterial catheter
* Patient with Radial Arterial Catheter Contraindication
* Radial arterial catheter placed by an anesthesiologist nurse student

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult who have an scheduled cardiac or aortic surgery at Montpellier University Hospital
Sampling Method: Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Failure to insert a radial artery catheter (KTA) by the nurse anesthesiologists | Day 1
  Failure to insert the radial KTA by the nurse anesthesiologist defined as follows: ≥ 3 punctures (by the nurse anesthetist) or need to change of doctor operator (nurse anesthesiologist to Anesthesiologist - Resuscitator) or change of puncture site (radial to radial contralateral or other site). All professionals involved are blinded to the echographic measures of the radial artery.

SECONDARY OUTCOMES:
Internal radial artery diameter | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
External radial artery diameter | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
Internal area of the radial artery | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
External area of the radial artery | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
Calcification of arterial wall (yes/no) | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
Thickness of arteria wall | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
Ratio between internal and external arteria diameter | Day 1
  Measured on echographic exam. Image acquisition done by an independent nurse anesthesist (not involved in the management of the same patient). Radial artery diameter measured on these images, later, by an anaesthesiologist-Resuscitator physician.
Clinical characteristics at baseline | Day 1
  Age, sex, body mass index, ASA score, duration of preoperative fasting, cardiovascular risk factors, cardiovascular conditions, wrist circumference, pulse force of the radial, ulnar, and brachial arteries (no pulse / feeble pulse / normal pulse), mean arterial pressure at punction time, dose of vasopressants (ephedrine, neosynephrine, noradrenaline) at punction time
Punction-related adverse events | 6 months
  Hematoma, dissection, thrombosis, ischemia, false aneuvrysm, infection, pain.
Duration of arterial punction | Day 1
  delay between first pulse palpation and end of bandage on a functional catheter
Duration of patient management | 28 days
  duration of anaesthesia, duration of presence in surgery room, length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme PANIEGO, Principal Investigator — University hospital of Montpellier, Montpellier, France, 34295
Locations (1):
- University hospital of Montpellier, Montpellier, France